CLINICAL TRIAL: NCT02072122
Title: The Influence of the Hormonal Fertility Treatment of Women, on the Eye Surface and the Eye Dryness
Brief Title: Estrogen and the Outer Eye in Women During Fertility Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: EOEDFT-2
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Dry Eye Syndromes
Keywords: dry eye; fertility treatment; Meibomian gland dysfunction; supra physiologic estrogen level
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples Without DNA — Blood tests (hormones level)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- women during fertility treatment

SUMMARY:
The purpose of this study is to determine the relation between estrogen and progesterone levels, and between dryness of the eyes, in women during their fertile years.

DETAILED DESCRIPTION:
Women during their fertility treatments will be submitted to the research. The research will include 3 meetings with a doctor from the ophthalmology department. Each meeting will be individual for each participant of the research.

The meetings will take place during the day of regular appointment of the participant to the fertility clinic.

Meeting #1:

During first visit to the fertility clinic for the stimulation process.

During this day will be done:

1.Submission of the patient to the research and signing on letter of agreement 2.Blood tests for estrogen, progesterone, luteinizing hormone (LH) 3.Eye examination: 3a. Filling of Schein Questionnaire 3b. Examination of the external eye: 1.microscope, 2.Schirmer test (paper strips inserted into the eye for several minutes to measure the production of tears), 3. tear break up time test (checking the eye with the fluorescein light after painting the eye with fluorescein dye) 3c. Checking the Intra Ocular Pressure with Tonometer

Meeting #2:

During visit to the fertility clinic for the egg collection (about 10 days after meeting #1)

During this day will be done:

1.Blood tests for estrogen, progesterone, luteinizing hormone (LH) 2.Eye examination: 2a. Filling of Schein Questionnaire 2b. Examination of the external eye: 1.microscope, 2.Schirmer test (paper strips inserted into the eye for several minutes to measure the production of tears), 3. tear break up time test (checking the eye with the fluorescein light after painting the eye with fluorescein dye) 2c. Checking the Intra Ocular Pressure with Tonometer

Meeting #3:

During visit to the fertility clinic for the pregnancy test (about 14 days after meeting #2)

During this day will be done:

1. Blood tests for estrogen, progesterone, luteinizing hormone (LH)
2. Eye examination:

2a. Filling of Schein Questionnaire 2b. Examination of the external eye: 1.microscope, 2.Schirmer test (paper strips inserted into the eye for several minutes to measure the production of tears), 3. tear break up time test (checking the eye with the fluorescein light after painting the eye with fluorescein dye) 2c. Checking the Intra Ocular Pressure with Tonometer

Collection and summary of all the data End of the research

ELIGIBILITY:
Inclusion Criteria:

* women during fertility treatment
* without any known eye diseases
* no current or past history of treatment against dry eye

Exclusion Criteria:

* known eye disease
* current or past history of treatment against dry eye

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: fertility clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Evidence of clinically definite dry eye confirmed by Schirmer test and tear break up time test | 24 days

SECONDARY OUTCOMES:
Evidence of clinically definite dry eye confirmed by Schirmer test and tear break up time test during each on of the meetings #1,#2 (day 0, day 10) | 0 days, 10 days